CLINICAL TRIAL: NCT00183872
Title: Phase II Study of Irinotecan and Docetaxel in Patients With Metastatic or Unresectable Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of Irinotecan and Docetaxel in Patients With Metastatic or Unresectable Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3G-03-5
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-12

CONDITIONS: Gastric Cancer; Esophageal Neoplasms
Keywords: Gastroesophageal cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Irinotecan; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 - Irinotecan and Docetaxel (Experimental): Irinotecan given day 1 and 8 every 21 days Docetaxel given day 1 and 8 every 21 days
  Interventions: Drug: irinotecan, docetaxel

INTERVENTIONS:
Drug: irinotecan, docetaxel — docetaxel 30 mg/m2 IV infusion days 1 and 8, with irinotecan 65 mg/m2 IV infusion on days 1 and 8.

SUMMARY:
This study is for people with advanced gastric or gastroesophageal cancer. This study is being done to find out how long it takes tumors to grow after receiving treatment with the drugs irinotecan (also known as CPT-11) and docetaxel (also known as Taxotere). Irinotecan is a drug that has been approved by the Food and Drug Administration (FDA). Irinotecan has been approved for treatment of cancer of the colon and rectum. Docetaxel is another drug approved by the FDA. Docetaxel is approved for treatment of breast, prostate and lung cancer. However, the FDA has authorized the use of irinotecan and docetaxel in this study. This study will evaluate the effects of these drugs on participant's tumors. The side effects of the combination of irinotecan and docetaxel will also be evaluated. This study will also measure the levels of certain substances in participant's tumors. These substances, called genes (which are the cell's blueprint), affect how people's bodies react to the cancer drugs. Genes will also be measured in participant's blood. The researchers want to see if these substances can predict response to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented unresectable or metastatic gastric cancer or gastroesophageal adenocarcinoma and histologic confirmation of the diagnosis with tumor.
* Patients must have received one prior chemotherapeutic regimen for metastatic or unresectable disease. Patients may not have received prior therapy with irinotecan or a taxane.
* Tissue from tumor must be available. This may be paraffin embedded tissue from previous biopsy/resection or if it is not available, a repeat biopsy must be performed.
* Patients must agree to have a 20 cc blood sample drawn in addition to routine labs with each cycle of chemotherapy.
* Patients must have measurable disease by clinical exam or radiologic studies, that is at least one lesion measurable in at least one dimension, measuring 10 mm or more on a spiral CT scan, or at least 20 mm by an exam or a non-spiral scan. If prior radiation therapy was administered, measurable disease must be outside the radiation field.
* Patients must have a Zubrod performance status of 0-2.
* Patients must have a predicted life expectancy of at least 12 weeks.
* Patients must have:

  * a pre-treatment granulocyte count (i.e., segmented neutrophils + bands) of >1,500/mm3,
  * a hemoglobin level of greater than or equal to 9.0 gm/dl, and
  * a platelet count of >100,000/mm3.
* Patients must have adequate renal function as documented by a calculated creatinine clearance > 60.
* Patients must have adequate hepatic function as documented by a serum bilirubin less than or equal to the institutional upper limit of normal, regardless of whether patients have liver involvement secondary to tumor.
* No major surgery within 1 month of starting study drug.
* Women of childbearing potential must have a negative pregnancy test.
* Peripheral neuropathy: must be < grade 1

Exclusion Criteria:

* Patients may not have a history of an allergy to irinotecan.
* Patients with any active or uncontrolled infection, including known HIV infection.
* Patients with psychiatric disorders that would interfere with consent or follow-up.
* Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy.
* Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on treatment and for at least 3 months thereafter.
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis.
* Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other anti-epileptic prophylaxis are ineligible.
* Patients with any other severe concurrent disease, which in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04-14 (Actual); Primary Completion 2014-10-20 (Actual); Study Completion 2015-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — University of Southern California (U.S.C.)/ Norris Comprehensive Cancer Center
Locations (1):
- University of Southern California (U.S.C.)/ Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University of Southern California cancer center facilities between April 14, 2005 and January 11, 2012.
Pre-assignment Details: There are no pre-assignment requirements for this study.
Period: Overall Study
Arm/Group | Arm 1 - Irinotecan and Docetaxel
Started | 40
Completed | 24
Not Completed | 16
Not completed — Death | 3
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 2
Not completed — Drug delayed more than 28 days | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 - Irinotecan and Docetaxel
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete, Partial, Stable and Progression)
Description: Objective response was defined using standard RECIST criteria. CR (complete response) = disappearance of all target lesions; PR (partial response) = 30% decrease in the sum of the longest diameter or target lesions; PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions SD (stable disease) = small changes that do not meet criteria of CR, PR, and PD.
Time Frame: every 2 cycles
Population: Population analyzed included all participants who received at least 6 weeks of treatment (or who were discontinued due to progressive disease or for reason of toxicity within the first 6 weeks of study). Two subjects had no tumor evaluation and follow up data available. Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Irinotecan and Docetaxel
Number analyzed (Participants) | 38
participants
  CR | 0
  PR | 7
  SD | 22
  PD | 9

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is measured from the start of treatment until the time the participant is first recorded as having disease progression, or death due to any cause. If a participant has not progressed or died, progression free survival is censored at the time of the last follow up.
Time Frame: every 2 cycles
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Irinotecan and Docetaxel
Number analyzed (Participants) | 38
Months | 4.1 [2.9 to 6]

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug is given
Description: Assessed from date on study until 30 days after last dose of drug is given. Assessment is based on CTCAE version 3.0.
Arm/Group | Arm 1 - Irinotecan and Docetaxel
All-Cause Mortality (participants affected / at risk) | 3/40
Serious Adverse Events (participants affected / at risk) | 29/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Irinotecan and Docetaxel (N=40)
Alkaline Phosphatase Increased (Investigations) | 1 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (2)
AST, SGOT (serum glutamic oxaloacestic transaminase) (Investigations) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 4 (8)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 (12)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (9)
Death not associated with CTCAE term (Death NOS) (General disorders) | 1 (1)
Death not associated with CTCAE term (Disease progression NOS) (General disorders) | 1 (1)
Death not associated with CTCAE term (Sudden death) (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (5)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)
Infection (Blood) (Infections and infestations) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC < 1.0 x 10e9/L
Dizziness (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain (Abodmen NOS) (Gastrointestinal disorders) | 2 (2)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Head/headache) (Nervous system disorders) | 2 (2)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 21 (61)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 9 (15)
Pain (Head/headache) (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (17)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Irinotecan and Docetaxel (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 36 (174)
Leukocytes (total WBC) (Investigations) | 11 (20)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 11 (33)
Platelets (Investigations) | 5 (9)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 27 (110)
Fever (General disorders) | 6 (7) — In the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L
Insomnia (Psychiatric disorders) | 10 (20)
Rigors/chills (General disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Weight loss (Investigations) | 11 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 27 (98)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (14)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (10)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 24 (63)
Constipation (Gastrointestinal disorders) | 10 (21)
Dehydration (Gastrointestinal disorders) | 9 (14)
Diarrhea (Gastrointestinal disorders) | 22 (54)
Mucositis/stomatitis (clinical exam (Oral cavity) (Gastrointestinal disorders) | 1 (2)
Mucositis/stomatitis (functional/symptomatic) (Oral cavity) (Gastrointestinal disorders) | 4 (8)
Nausea (Gastrointestinal disorders) | 22 (69)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (42)
Hemorrhage, pulmonary/upper respiratory (Nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: limb (General disorders) | 11 (16)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 15 (42)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 16 (50)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (4)
Alkaline Phosphatase (Investigations) | 21 (65)
Bilirubin (Investigations) | 4 (7)
Calcium,serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (3)
Creatinine (Investigations) | 3 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (25)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (4)
Confusion (Psychiatric disorders) | 1 (2)
Dizziness (Nervous system disorders) | 6 (8)
Mood alteration (Depression) (Psychiatric disorders) | 2 (4)
Neuropathy (Nervous system disorders) | 24 (98)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (2)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes